CLINICAL TRIAL: NCT02152228
Title: A Pilot Study to Assess the Safety and Efficacy of Oral PTH (1-34) in the Treatment of Hypoparathyroidism
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Entera Bio Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ENT-03-2014
Record Dates: First submitted 2014-04-22; First posted 2014-06-02 (Estimated); Last update posted 2015-10-07 (Estimated); Status verified 2015-10

CONDITIONS: Hypoparathyroidism
MeSH Terms: conditions — Hypoparathyroidism | interventions — Teriparatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Oral Parathyroid Hormone (1-34) (Experimental): Oral administration of EnteraBio's Oral Parathyroid Hormone (1-34)
  Interventions: Drug: EnteraBio's Oral Parathyroid Hormone (1-34)

INTERVENTIONS:
Drug: EnteraBio's Oral Parathyroid Hormone (1-34) — Oral administration
  Other Names: Teriparatide

SUMMARY:
This is an observational, international, open label, pilot study to evaluate the safety, tolerability and efficacy of an oral PTH (1-34) preparation produced by Entera Bio in adult hypoparathyroid volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of primary hypoparathyroidism for more than 1 year.
* Currently taking >1.0 grams of Calcium/day with a correlate alpha D3 dose.
* 25(OH)D levels ≥ 20 ng/ml.
* Signed informed consent.
* BMI 18 - 30 kg/m2, inclusive.
* Full blood count should be within the reference range as per WHO criteria. Minor abnormalities will be assessed by the Principle Investigator and after discussion with sponsor patients may still be entered if these are felt to be of "no clinical importance". Abnormalities due to hypoparathyroidism related are acceptable and will not constitute exclusion.
* Patients with significant liver function impairment (liver enzymes above x3 the upper limit of normal range as per WHO criteria) will be excluded.
* Subjects able to adhere to the visit schedule and protocol requirements.

Exclusion Criteria:

* Haemoglobin <12 g/dL (females)/ <13gm/dL (males) [lower limit of reference range 12-15 & 13-17]
* Impaired renal function
* impaired liver function; ALT >38 international units per liter (IU/L), or ALP>125 IU/L
* Significant drug or alcohol abuse as assessed by the Principal Investigator
* Allergy to soy bean products
* Presence of kidney or urinary tract stones
* Concurrent therapy that, in the Investigator's opinion, would interfere with the evaluation of the safety or efficacy of the study medication.
* Treatment with any investigational product within the last 30 days, enrollment or intention to enroll in any active study involving the use of investigational devices or drugs.
* Presence of any other condition or circumstance that, in the judgment of the Investigator, might increase the risk to the patient or decrease the chance of obtaining satisfactory data to achieve the objectives of the study.
* Active infections
* Pregnancy or suspected pregnancy. Female subjects must have a negative serum pregnancy test at screening and be willing and able to use a medically acceptable method of birth control (reliable use of oral contraceptive, non-hormonal intrauterine device with condom, or diaphragm with condom, or condom with spermicide) from the screening visit through the study termination visit or declare that they are abstaining from sexual intercourse from the screening visit through the study termination visit or are surgically sterile (have undergone bilateral tubal ligation, bilateral oophorectomy, or hysterectomy) or post-menopausal. Postmenopausal women are defined as women with menstruation cessation for 12 consecutive months prior to signing of the informed consent form.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-07; Primary Completion 2015-06 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | up to 17 weeks
  safety will be measured by monitoring and recording adverse events related to hyper- and hypocalcemia
Reduction in use of exogenous calcium supplement and/or alpha D3 supplement | up to 17 weeks
Tolerability- The rate of discontinuation of patients' participation in the study due to adverse events | up to 17 weeks
Plasma calcium levels | at baseline and 60 minutes post-dose
Peak Plasma Concentration (Cmax)of treatment | at baseline and time-points post-dose
  To study the pharmacokinetic profile of PTH absorption

SECONDARY OUTCOMES:
The volunteers' compliance to treatment | up to 17 weeks
  Compliance to treatment defined as proportion taking >80% study medication (good), 60-80% (satisfactory) and <60% (poor)
Patient quality of life | up to 17 weeks
  Patients will report a Quality Of Life (QOL) review

CONTACTS AND LOCATIONS:
Overall Officials: Sophia Ish Shalom, MD, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Lin Medical Center, Haifa, Israel